CLINICAL TRIAL: NCT01237340
Title: A Phase IIIb, Open-label, Single-arm, Multicenter Study to Assess the Immunogenicity of the Recombinant-Human Growth Hormone (r-hGH) Liquid Multidose Formulation (Saizen® Solution for Injection) When Administered to Male and Female Adults With Documented Growth Hormone Deficiency (GHD)
Brief Title: Saizen® Solution for Injection Adult Growth Hormone Deficiency (GHD) Immunogenicity Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor voluntarily terminated this trial because compliance to strict Good Clinical Practice (GCP) requirements was not ensured - No safety concerns
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 701048-009
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Growth Hormone Deficiency (GHD)
Keywords: Adult Growth Hormone Deficiency (AGHD); immunogenicity; growth hormone; antibodies; GH biomarkers; IGF-I
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Saizen® (Experimental)
  Interventions: Drug: Saizen®

INTERVENTIONS:
Drug: Saizen® — Single dose of Saizen® (recombinant human growth hormone, r-hGH) solution for injection will be administered subcutaneously for 26 weeks. Dosage regimen will be in accordance with marketed formulation of Saizen® (freeze-dried formulation), based on locally approved product labeling.
  Other Names: r-hGH; Somatropin

SUMMARY:
To assess the immunogenicity of Saizen® solution for injection in adult subjects with documented Growth Hormone Deficiency (GHD).

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects, 18-60 years of age, inclusive, at the time the informed consent is signed
* Subjects who have confirmed adult GHD
* Subjects who are growth hormone (GH) treatment-naive or had received Saizen® (freeze-dried formulation) for pediatric GHD (PGHD), or are currently receiving Saizen® freeze-dried formulation for adult GHD (AGHD)
* Subjects who have binding antibody-negative (BAbs-) at screening
* Subjects who have no evidence of concomitant disease, intercurrent illness, or resultant therapy that would interfere with subject compliance, the evaluation of study results, or compromise the safety of the subject
* Female subjects of childbearing potential who have a negative serum pregnancy test at the screening visit (and at each scheduled visit during the study)
* Subjects who are willing to comply with the procedures of the study
* Subjects who are willing to sign an Independent Ethics Committee/Institutional Review Board approved informed consent form
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Subjects who are currently receiving or have previously received treatment for adult GHD or any other indication, including PGHD, with a commercial GH product other than Saizen® freeze-dried formulation
* Subjects who had a chronic underlying disease within 6 months prior to screening or concomitant medication(s) that in the opinion of the investigator would exclude the subject from the trial
* Subjects who have significant renal impairment
* Subjects who have diabetes mellitus
* Subjects who are immunosuppressed
* Subjects who have a current malignancy or a history of any malignancy (excluding fully-treated basal cell carcinoma)
* Subjects who have participated in another study and received an investigational drug within 30 days prior to screening visit
* Subjects who have clinically significant abnormal laboratory value(s)
* Subjects who have known hypersensitivity or allergy to exogenous human GH or any of the excipients or phenol, the bacteriostatic agent in the Saizen® solution for injection
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.A., Geneva
Locations (1):
- US Medical Information, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saizen®
Started | 59
Completed | 19
Not Completed | 40
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Early termination of the trial | 36

BASELINE CHARACTERISTICS:
Arm/Group | Saizen®
Number analyzed (Participants) | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 44.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Positive Binding Antibodies (BAbs+) to Saizen®
Description: Binding antibodies (BAbs) are all antibodies which are capable of binding to the investigational drug molecule (Saizen®), irrespective of their binding site.
Time Frame: Baseline up to Week 26
Population: Modified Intent-to-Treat (MITT) population consisted of all the participants who received at least 1 dose of study medication and had at least one post-baseline BAbs assessment.
Measure: Number; unit: participants
Arm/Group | Saizen®
Number analyzed (Participants) | 59
participants | 1

2. Secondary Outcome: Number of Participants Who Developed Positive Neutralizing Antibodies (NAbs+) to Saizen®
Description: Neutralizing antibodies (NAbs) are defined as a subgroup of BAbs which bind to the active sites of the investigational drug molecule (Saizen®) and therefore neutralize its potency.
Time Frame: Baseline up to Week 26
Population: MITT population consisted of all the participants who received at least 1 dose of study medication and had at least one post-baseline BAbs assessment.
Measure: Number; unit: participants
Arm/Group | Saizen®
Number analyzed (Participants) | 59
participants | 0

3. Secondary Outcome: Insulin-like Growth Factor-I (IGF-1) Levels
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 13, Week 18, Week 26
Population: Safety population consisted of all the participants who received at least 1 dose of study medication and had at least one post-baseline safety assessment. 'N' (number of participants analyzed) = participants who were evaluated for this measure and "n"= participants who were analyzed at that particular time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: nanomole per liter (nmol/L)
Groups:
- GH Treatment-Naive: Growth hormone (GH) Treatment-Naive participants were those who did not receive any prior treatment with Saizen® before initiation of the trial. Single dose of Saizen® (recombinant human growth hormone, r-hGH) solution for injection will be administered subcutaneously for 26 weeks. Dosage regimen will be in accordance with marketed formulation of Saizen® (freeze-dried formulation), based on locally approved product labeling.
- GH Treatment-Experienced: Growth hormone (GH) Treatment-experienced participants were those who had undergone treatment with the freeze-dried formulation of Saizen® before initiation of the trial. Growth hormone (GH) Treatment-experienced participants were those who had undergone treatment with the freeze-dried formulation of Saizen® before initiation of the trial. Single dose of Saizen® (recombinant human growth hormone, r-hGH) solution for injection will be administered subcutaneously for 26 weeks. Dosage regimen will be in accordance with marketed formulation of Saizen® (freeze-dried formulation), based on locally approved product labeling.
Arm/Group | GH Treatment-Naive | GH Treatment-Experienced
Number analyzed (Participants) | 49 | 8
nanomole per liter (nmol/L)
  Baseline (n = 49, 8) | 11.492 (6.694) | 20.225 (10.194)
  Week 2 (n = 47, 8) | 18.923 (10.394) | 28.663 (9.001)
  Week 4 (n = 49, 8) | 19.914 (11.532) | 24.500 (11.176)
  Week 8 (n = 49, 8) | 21.155 (10.520) | 27.075 (6.815)
  Week 13 (n = 46, 8) | 23.415 (8.020) | 26.413 (8.767)
  Week 18 (n = 31, 4) | 24.948 (9.300) | 25.650 (8.502)
  Week 26 (n = 48, 8) | 24.117 (11.085) | 27.438 (12.402)

4. Secondary Outcome: Insulin-like Growth Factor-I Standard Deviation Score (IGF-1 SDS)
Description: Insulin-like Growth Factor-1 Standard Deviation Score (IGF-1 SDS) was provided by the central laboratory; its calculation is based on the actual value of IGF-1 minus mean reference value of IGF-1 divided by reference standard deviation of IGF-1.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 13, Week 18, Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: standard deviation score
Groups:
- GH Treatment-Experienced: Growth hormone (GH) Treatment-experienced participants were those who had undergone treatment with the freeze-dried formulation of Saizen® before initiation of the trial. Single dose of Saizen® (recombinant human growth hormone, r-hGH) solution for injection will be administered subcutaneously for 26 weeks. Dosage regimen will be in accordance with marketed formulation of Saizen® (freeze-dried formulation), based on locally approved product labeling.
Arm/Group | GH Treatment-Naive | GH Treatment-Experienced
Number analyzed (Participants) | 49 | 8
standard deviation score
  Baseline (n = 49, 8) | -2.914 (2.268) | -0.550 (2.274)
  Week 2 (n = 47, 8) | -0.926 (2.300) | 0.951 (1.411)
  Week 4 (n = 49, 8) | -0.867 (2.615) | 0.153 (1.762)
  Week 8 (n = 49, 8) | -0.464 (2.274) | 0.834 (1.063)
  Week 13 (n = 46, 8) | 0.212 (1.832) | 0.666 (1.225)
  Week 18 (n = 31, 4) | 0.455 (1.816) | 1.043 (1.144)
  Week 26 (n = 48, 8) | 0.167 (2.016) | 0.544 (1.894)

5. Secondary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 13, Week 18, Week 26
Population: Safety population consisted of all the participants who received at least 1 dose of study medication and had at least one post-baseline safety assessment. Here "n" signifies number of participants analyzed at that particular time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GH Treatment-Naive | GH Treatment-Experienced
Number analyzed (Participants) | 51 | 8
nmol/L
  Baseline (n = 51, 8) | 124.941 (31.899) | 133.375 (36.024)
  Week 2 (n = 49, 8) | 137.408 (35.088) | 162.125 (35.203)
  Week 4 (n = 49, 8) | 144.592 (32.632) | 147.750 (26.451)
  Week 8 (n = 50, 8) | 147.460 (36.381) | 156.625 (36.190)
  Week 13 (n = 47, 8) | 149.404 (28.272) | 151.875 (35.679)
  Week 18 (n = 32, 4) | 148.813 (39.754) | 155.500 (36.235)
  Week 26 (n = 49, 8) | 152.429 (35.649) | 147.500 (30.402)

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs): Any untoward medical occurrence in the form of signs, clinically significant abnormalities in laboratory findings, diseases, symptoms, or worsening of complications. TEAEs: AEs occurring after the first administration of Saizen® solution for injection (on Day 1) up to the scheduled routine post treatment follow-up visit (4 weeks [28 days] after the final administration of Saizen® solution for injection).
Time Frame: Day 1 up to 28 days after last dose of study treatment
Population: Safety population consisted of all the participants who received at least 1 dose of study medication and had at least one post-baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Saizen®
Number analyzed (Participants) | 59
participants | 40

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of study treatment
Description: TEAEs: AEs occurring after the first administration of Saizen® solution for injection (on Day 1) up to the scheduled routine post treatment follow-up visit (4 weeks [28 days] after the final administration of Saizen® solution for injection).
Arm/Group | Saizen®
Serious Adverse Events (participants affected / at risk) | 3/59
Other Adverse Events (participants affected / at risk) | 13/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen® (N=59)
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen® (N=59)
Oedema peripheral (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 4
Headache (Nervous system disorders) | 3
Insulin-like growth factor increased (Investigations) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other